CLINICAL TRIAL: NCT00892203
Title: A Multi-centre, Randomized, Double-blind, Parallel Group, Active and Placebo Controlled, Proof of Concept Study in Patients With Acute Migraine to Assess the Efficacy, Safety and Tolerability of Single Oral Doses of BGG492
Brief Title: Efficacy and Safety of BGG492 in the Treatment of Migraine
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CBGG492A2204; 2008-005392-10 (EudraCT Number)
Record Dates: First submitted 2009-05-01; First posted 2009-05-04 (Estimated); Last update posted 2020-12-17 (Actual); Status verified 2016-03

CONDITIONS: Migraine
Keywords: Migraine; Headache
MeSH Terms: conditions — Migraine Disorders; Headache | interventions — selurampanel; Sumatriptan

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Active (Experimental)
  Interventions: Drug: BGG492
- Comparator (Active Comparator)
  Interventions: Drug: Sumatriptan
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: BGG492
  Arms: Active
Drug: Sumatriptan
  Arms: Comparator
Drug: Placebo
  Arms: Placebo

SUMMARY:
This study will assess the efficacy and safety of BGG492 used to treat migraine pain.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of moderate to severe migraine for at least 1 year
* At least 1 migraine episode, but not more 15 migraine days per month
* Past use of triptans
* Migraine onset before 50 years of age

Exclusion Criteria:

* Diagnosis of basilar, ophthalmoplegic or hemiplegic migraine.
* More than 6 non-migraine headaches per month
* Patients receiving migraine prophylaxis treatment
* Patients receiving regular treatment with psychoactive drugs
* Smokers
* Patients with a very high or low body weight Other protocol-defined inclusion/exclusion criteria may apply

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 75 (Actual)
Dates: Start 2009-04; Primary Completion 2010-08 (Actual); Study Completion 2010-08 (Actual)

PRIMARY OUTCOMES:
Reduction in migraine pain | 2 hours

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Investigator Site
Locations (13):
- United States (2):
  - California Clinical Trials, 1560 Chevy Chase Drive, Suite 140, Glendale, California
  - California Clinical Trials, 15625 Lakewood Boulevard, Paramount, California
- Germany (10):
  - Novartis Investigative Site, Berlin
  - Novartis Investigative Site, Essen
  - Novartis Investigative Site, Göttingen
  - Novartis Investigator Site, Hamburg
  - Novartis Investigative Site, Kiel
  - Novartis Investigative Site, Königstein
  - Novartis Investigative Site, Munich
  - Novartis Investigator Site, Munich
  - Novartis Investigative Site, Münster
  - Novartis Investigative Site, Würzburg
- Novartis Investigative Site, Barcelona, Spain

REFERENCES:
- [Derived] Gomez-Mancilla B, Brand R, Jurgens TP, Gobel H, Sommer C, Straube A, Evers S, Sommer M, Campos V, Kalkman HO, Hariry S, Pezous N, Johns D, Diener HC; BGG492 Study Group. Randomized, multicenter trial to assess the efficacy, safety and tolerability of a single dose of a novel AMPA receptor antagonist BGG492 for the treatment of acute migraine attacks. Cephalalgia. 2014 Feb;34(2):103-13. doi: 10.1177/0333102413499648. Epub 2013 Aug 20. PMID 23963355
- See also: Results for CBGG492A2204 from the Novartis Clinical Trials website — https://www.novctrd.com/ctrdweb/trialresult/trialresults/pdf?trialResultId=5409